CLINICAL TRIAL: NCT03459066
Title: Predictive Factors and Time of Onset of Spasticity in Post-stroke Patients and Their Relationship With the Functionality and Quality of Life.
Brief Title: Predictors Factors and Time of Onset of Spasticity and Their Relationship With the Functionality and Quality of Life.
Status: Completed | Type: Observational
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, ARLETTE PATRICIA DOUSSOULIN SANHUEZA, Dr. Arlette Doussoulin, Universidad de La Frontera
Other Study IDs: Spasticity Factors
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Post Stroke Spasticity
Keywords: Spasticity; Stroke; Predictors; Functionality; Quality of life
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Institution-Group 8 district: Group of patients belonging to institutions of district 8. Patients will be evaluated in 3 different times with different assessment instruments for tone, functionality and quality of life.
  Interventions: Diagnostic Test: Institution-Group
- Institution-Group 9 district: Group of patients belonging to institutions of district 9. Patients will be evaluated in 3 different times with different assessment instruments for tone, functionality and quality of life.
  Interventions: Diagnostic Test: Institution-Group
- Institution-Group 10 district: Group of patients belonging to institutions of district 10. Patients will be evaluated in 3 different times with different assessment instruments for tone, functionality and quality of life.
  Interventions: Diagnostic Test: Institution-Group

INTERVENTIONS:
Diagnostic Test: Institution-Group — The study includes three measurement times:
  * Time 1 (T1): corresponds to the first measurement, which will take place between the 3rd and 10th day of hospitalization.
  * Time 2 (T2): corresponds to the second measurement, which will be carried out 3 months after the first measurement.
  * Time 3 (T3): corresponds to the third measurement, which will be carried out 12 months after the first measurement.
  The evaluations will be tone, functionality and quality of life.

SUMMARY:
Spasticity is part of the syndrome motor neuron following a Stroke. It is a clinical sign of great complexity that generates disability, limiting the function and altering the quality of life of the subjects, generating great impact on families and society.

Identify times and characteristics of appearance; as well as its predictive factors can support an early intervention, orienting and strengthening the work of the rehabilitation team.

Determine the times of establishment, location and factors that favor the development of spasticity in acute stage and how it influences the functionality, quality of life and emotional level of post-stroke patients in hospital facilities.

Through this proposal, it is proposed to generate a new line of research that allows the development of scientific evidence in the area of neurorehabilitation, specifically in the field of spasticity, through the identification of establishment times, affected structures and predominant patterns in the extremities; as well as determining factors that favor the development of spasticity and its impact on post-stroke functionality and quality of life.

This information will strengthen the rehabilitative process of these subjects and the actions of the rehabilitation team, supporting the identification of preventive measures and implementing effective interventions that allow achieving better motor and functional results, in search of an optimal recovery.

DETAILED DESCRIPTION:
A correlational (non-experimental), longitudinal, prospective follow-up design will be used for descriptive and predictive purposes.

The sample will consist of 150 subjects who meet the inclusion criteria, sign the informed consent and who will be treated during the year 2018 at the Hospital and the Clinic.

The study will include three measurement times: Time 1, during the first 10 days of hospitalization (T1); Time 2, at 3 months after T1; and Time 3, at 12 months after T1.

At each time of measurement, the study variables will be evaluated by 4 professionals trained in the following instruments: the Ashworth Scale to assess spasticity; To measure global functionality, the Barthel Index will be applied and, to assess functionality of the upper extremity, the Action Research Arm scale will be used; The Quality of Life Scale for Stroke-38 will be used to assess quality of life and emotional level. In addition, in time 1 the sociodemographic and clinical characteristics of the sample will be evaluated through a clinical record prepared for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Have an age between 20 and 80 years, with no previous history of motor disability.
* Being hospitalized with a diagnosis of ischemic or hemorrhagic stroke in the acute period.
* Present a history with a single stroke event confirmed by Computerized Axial Tomography.
* Without severe cognitive commitment, that is, score greater than 14 on the MiniMental Abbreviated scale.
* Stable hemodynamically.
* Voluntarily accept participation in the study through the signing of informed consent, either personally or through a family member.

Exclusion Criteria:

* Present sensitive aphasia.
* Have a medical contraindication.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will be constituted by all the subjects with a medical diagnosis of stroke in the acute phase, attended during 2018 at the Dr. Hernán Henríquez Aravena Hospital and the Alemana Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Ashworth Scale | 6 months
  Instrument used in the assessment of spasticity. Graduates the tone from 0 (no increase in tone) to 4 (rigid extremity in flexion or extension), it is based on the examiner manually moving a limb of the patient, in the whole of the possible joint range (in the clinical setting it is use 1 second to perform the complete joint travel) and perceive the resistance that a muscle offers when stretched.
Action Research Arm | 6 months
  This Instrument was constructed to determine the functional recovery of the upper limb. It is composed of 19 items grouped in 4 subtest, including each subtest: 6 items of grip, 4 items taken, 6 items of clip, 3 items of thick movement. All the items are evaluated with a scale of 4 points from 0 to 3, where 0 represents no movement and 3 normal movement for the task.
Barthel Index | 6 months
  Scale that assesses the level of patient independence with respect to performing Activity Daily Life. The values assigned to each activity depend on the time spent and help to carry it out.
  The activities are valued differently, being able to assign 0, 5, 10 or 15 points. The global range can vary between 0, completely dependent, and 100 points, completely independent.

CONTACTS AND LOCATIONS:
Overall Officials: Arlette Doussoulin, PhD, Principal Investigator — Universidad de La Frontera
Locations (1):
- Universidad de La Frontera, Temuco, Chile

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided this item.